CLINICAL TRIAL: NCT01356992
Title: A Multicenter, Randomized, Open-label, Non-inferiority Phase III Study, Between Low-Molecular Weight Heparins, Versa® (Enoxaparin - Eurofarma) and Clexane® (Enoxaparin - Sanofi-Aventis), in Patients With High-risk Acute Coronary Syndrome Without ST-segment Elevation.
Brief Title: Patients With High-risk Acute Coronary Syndrome Without ST-segment Elevation
Acronym: VECOR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change in strategy regarding the product by the company
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 117
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Non ST Segment Elevation Myocardial Infarction; Unstable Angina
Keywords: non-inferiority phase III study; Low-Molecular Weight Heparin; Versa® (enoxaparin - Eurofarma); Clexane® (enoxaparin - Sanofi-Aventis); Acute coronary syndrome without ST-segment elevation
MeSH Terms: conditions — Angina, Unstable | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clexane® (enoxaparin - Sanofi) (Active Comparator)
  Interventions: Drug: Enoxaparin
- Versa® (enoxaparin - Eurofarma) (Experimental)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Drugs will be provided by the sponsor to the study's patients on the reference presentation: 40 mg/0.4mL, 60 mg/0.6 mL and 80 mg/0.8 mL (solution for injection of enoxaparin sodium, 1 mg/ kg Sanofi-Aventis) or Eurofarma enoxaparin sodium (1 mg/ kg). The patients will use the drug corresponding to the arm of the study to which they were allocated. The drug administration must be performed through subcutaneous via on the dose of 1 mg/kg every 12 hours for at least 2 days and kept until the patient is discharged.

SUMMARY:
This non-inferiority study aims at comparing Versa® to the reference enoxaparin (Clexane®, Sanofi-Aventis) in patients with high-risk unstable angina and NSTEMI. The main justification is the search for scientific evidence to prove the Versa® effectiveness for this new therapeutic indication, since it is a product with potential for reducing costs, with effectiveness and safety comparable to the reference drug.

DETAILED DESCRIPTION:
To be included in this study, the eligible patients must meet all criteria below:

IC signature; The research subject must agree about following all instructions and perform the procedures and study visits; Men and women over the age of 18 and below the age of 75; History of angina of rest with a minimum duration of 20 minutes in the last 24 hours at the beginning and at least for 10 days.

Patient Randomization up to 6 hours after the arrival at the emergency sector.

Evidence of NSTEMI or unstable angina due to one or more of the following criteria:

1. Dynamic alterations on the T-wave (ST-segment depression or elevation > 1 mm, and/or T-wave inversions which are solved at least partially when the symptoms are relieved) or 2. Unevenly ST-segment (depression or elevation) in a transitional way under continuous derivations (V1+V2 or V3+V4 or V5+V6 or D1+AVL or D2+D3+AVF) or 3. Biochemical alteration on the myocardial necrosis markers (CKMB mass, troponin T or I and CPK), with the appearance of enzymatic curve, characterizing myocardial injury or 5. Pulmonary Edema; or 6. Angina associated to murmur of mitral regurgitation; or 7. Angina with heart sound to cardiac auscultation or throes; or 8. Angina with hypotension;

The patients who meet anyone of the criteria below will not be eligible for the study:

12-derivation-ECG with persistent ST-segment elevation; Diagnosis of angina by secondary cause (e.g., anemia, fever, hypovolemia, dehydration, use of cocaine); Use of non-fractionated heparin or low-molecular weight heparin in the prior 48 to the randomization; Concomitant diseases, such as severe renal failure (creatinine clearance lower than 30ml/min.) and hepatic, or other significant comorbidities under investigator judgment; Recent hemorrhagic cerebrovascular accident (last 12 months); Patient scheduled for cardiac surgery of myocardial revascularization; Use of drugs, alcohol abuse; Pregnancy or lactation; Recent neurosurgery or ophthalmic surgery (last 3 months); History or diagnosis of coagulopathy; Medical record containing allergy, hypersensibility or intolerance to any of the drug components to be used on this study, which is judged as clinically significant in the main investigator's opinion; Recent participation (last 12 months) in a clinical study.

ELIGIBILITY:
Inclusion Criteria:

* ICF signature;
* The research subject must agree about following all instructions and perform the procedures and study visits;
* Men and women over the age of 18 and below the age of 75;
* History of angina of rest with a minimum duration of 20 minutes in the last 24 hours at the beginning and at least for 10 days.
* Patient Randomization up to 6 hours after the arrival at the emergency sector.
* Evidence of NSTEMI or unstable angina due to one or more of the following criteria:

  1. Dynamic alterations on the T-wave (ST-segment depression or elevation > 1 mm, and/or T-wave inversions which are solved at least partially when the symptoms are relieved) or 2. Unevenly ST-segment (depression or elevation) in a transitional way under continuous derivations (V1+V2 or V3+V4 or V5+V6 or D1+AVL or D2+D3+AVF) or 3. Biochemical alteration on the myocardial necrosis markers (CKMB mass, troponin T or I and CPK), with the appearance of enzymatic curve, characterizing myocardial injury or 5. Pulmonary Edema; or 6. Angina associated to murmur of mitral regurgitation; or 7. Angina with heart sound to cardiac auscultation or throes; or 8. Angina with hypotension;

Exclusion Criteria:

* 12-derivation-ECG with persistent ST-segment elevation;
* Diagnosis of angina by secondary cause (e.g., anemia, fever, hypovolemia, dehydration, use of cocaine);
* Use of non-fractionated heparin or low-molecular weight heparin in the prior 48 to the randomization;
* Concomitant diseases, such as severe renal failure (creatinine clearance lower than 30ml/min.) and hepatic, or other significant comorbidities under investigator judgment;
* Recent hemorrhagic cerebrovascular accident (last 12 months);
* Patient scheduled for cardiac surgery of myocardial revascularization;
* Use of drugs, alcohol abuse;
* Pregnancy or lactation;
* Recent neurosurgery or ophthalmic surgery (last 3 months);
* History or diagnosis of coagulopathy;
* Medical record containing allergy, hypersensibility or intolerance to any of the drug components to be used on this study, which is judged as clinically significant in the main investigator's opinion;
* Recent participation (last 12 months) in a clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Frequency of death and infarction within 30 days after the admission in emergency | 30 days after the admission in emergency
  The study primary objective aims at evaluating the enoparaxin sodium (Eurofarma) effectiveness and safety on the treatment of patients with NSTE-ACS and high-risk ones, regarding the Sanofi-Aventis enoxaparin sodium. The primary endpoint will be the frequency of death and infarction within 30 days after the admission in emergency.

SECONDARY OUTCOMES:
Comparing the effectiveness and safety of the two formulations in patients with NSTE-ACS and high-risk ones | 30 days after the admission in emergency
  The secondary endpoints considered for the study are:
  Negative endpoints associated to ACS (shock, pulmonary congestion, arrhythmias, congestive heart failure, hemodynamic instability and reinfarction) during 30 days after the beginning of the treatment.
  Frequency of coronary angioplasty or surgical revascularization procedures; Rate of major bleeding during hospitalization according to TIMI criteria ; Incidence of hemotransfusion in the 30 days after the inclusion on the study.

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Salvador, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - São Jose Do Rio Preto, São Paulo
  - São Paulo, São Paulo